CLINICAL TRIAL: NCT02556788
Title: A Multi-Center, Randomized, Double-Blind, Parallel-Group Vehicle Controlled Study To Compare The Efficacy And Safety Of CD5789 (Trifarotene) 50µg/g Cream Versus Vehicle Cream In Subjects With Acne Vulgaris
Brief Title: Double-Blind Efficacy and Safety of CD5789 (Trifarotene) 50µg/g Cream Versus Vehicle Cream in Acne Vulgaris
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RD.06.SPR.18252
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Results first posted 2019-09-03 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2018-07

CONDITIONS: Acne Vulgaris
Keywords: Efficacy; Safety; Acne vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — trifarotene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CD5789 (Trifarotene) 50µg/g Cream (Experimental): CD5789 (trifarotene) 50µg/g Cream
  Interventions: Drug: CD5789 (trifarotene) 50µg/g Cream
- Placebo Cream (Placebo Comparator): Placebo Cream
  Interventions: Drug: Placebo Cream

INTERVENTIONS:
Drug: CD5789 (trifarotene) 50µg/g Cream — CD5789 (Trifarotene) 50µg/g cream applied once daily during 12 weeks.
  Arms: CD5789 (Trifarotene) 50µg/g Cream
Drug: Placebo Cream — Placebo cream applied once daily during 12 weeks.
  Arms: Placebo Cream

SUMMARY:
Assessment of the efficacy and safety of CD5789 (Trifarotene) 50µg/g cream applied once daily for 12 weeks in subjects with acne vulgaris.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a male or female, 9 years of age or older, at Screening visit.
* The Subject has moderate acne at Screening and Baseline.
* The subject is a female of non childbearing potential
* The subject is a female of childbearing potential with a negative pregnancy test and who is strictly abstinent or who agrees to use an effective and approved contraceptive method for the duration of the study and at least 1 month after the last study drug application.

Exclusion Criteria:

* The subject has severe forms of acne (e.g., acne conglobate, acne fulminant) or secondary acne form (e.g.,chloracne, drug-induced acne, etc.).
* The subject has any uncontrolled or serious disease or any medical or surgical condition that may either interfere with the interpretation of the trial results and/or put the subject at significant risk (according to the Investigator's judgment) if the subject takes part to the trial.
* The subject has been exposed to excessive ultraviolet (UV) radiation within one month prior to the Baseline visit or the subject is planning intense UV exposure during the study (i.e., occupational exposure to the sun, sunbathing, tanning salon use, phototherapy, etc.)
* The subject is unwilling to refrain from use of prohibited medication during the clinical trial

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1212 (Actual)
Dates: Start 2015-11; Primary Completion 2017-02-07 (Actual); Study Completion 2017-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Chan, Study Director — Galderma R&D
Locations (69):
- United States (29):
  - Galderma Investigational Site, Birmingham, Alabama
  - Galderma Investigational Site, Phoenix, Arizona
  - Galderma Investigational Site, Tucson, Arizona
  - Galderma Investigational Site, Fort Smith, Arkansas
  - Galderma Investigational Site, Los Angeles, California
  - Galderma Investigational Site, Murrieta, California
  - Galderma Investigational Site, Santa Ana, California
  - Galderma Investigational Site, Aventura, Florida
  - Galderma Investigational Site, Miami, Florida
  - Galderma Investigational Site, Miami Lakes, Florida
  - Galderma Investigational Site, West Palm Beach, Florida
  - Galderma Investigational Site, Corbin, Kentucky
  - Galderma Investigational Site, Beverly, Massachusetts
  - Galderma Investigational Site, Ann Arbor, Michigan
  - Galderma Investigational Site, Detroit, Michigan
  - Galderma Investigational Site, Brooklyn, New York
  - Galderma Investigational Site, Stony Brook, New York
  - Galderma Investigational Site, Wilmington, North Carolina
  - Galderma Investigational Site, Fort Washington, Pennsylvania
  - Galderma Investigational Site, Philadelphia, Pennsylvania
  - Galderma Investigational Site, Greer, South Carolina
  - Galderma Investigational Site, Goodlettsville, Tennessee
  - Galderma Invetsigational site, Austin, Texas
  - Galderma Investigational Site, Dallas, Texas
  - Galderma Investigational Site, Houston, Texas
  - Galderma Investigational Site, Pflugerville, Texas
  - Galderma Investigational Site, San Antonio, Texas
  - Galderma Investigational Site, Webster, Texas
  - Galderma Investigational Site, Walla Walla, Washington
- Czechia (6):
  - Galderma Investigational Site, Chomutov
  - Galderma Investigational Site, Hradec Králové
  - Galderma Investigational Site, Kutná Hora
  - Galderma Investigational Site, Olomouc
  - Galderma Investigational Site, Pardubice
  - Galderma Investigational Site, Prague
- Hungary (6):
  - Galderma Investigational Site, Budapest
  - Galderma Investigational Site, Debrecen
  - Galderma Investigational Site, Miskolc
  - Galderma Investigational Site, Pécs
  - Galderma Investigational Site, Szeged
  - Galderma Investigational Site, Szolnok
- Poland (9):
  - Galderma Investigational Site, Bialystok
  - Galderma Investigational Site, Gdansk
  - Galderma Investigational Site, Katowice
  - Galderma investigational Site, Katowice
  - Galderma Investigational Site, Lodz
  - Galderma Investigational Site, Sochaczew
  - Galderma Investigational Site, Warsaw
  - Galderma investigational Site, Warsaw
  - Galderma Investigational Site, Wroclaw
- Romania (4):
  - Galderma Investigational Site, Brasov
  - Galderma Investigational Site, Craiova
  - Galderma Investigational Site, Iași
  - Galderma Investigational Site, Târgu Mureş
- Russia (5):
  - Galderma Investigational Site, Krasnodar
  - Galderma Investigational Site, Lipetsk
  - Galderma Investigational Site, Moscow
  - Galderma Investigational Site, Saint Petersburg
  - Galderma Investigational Site, Sr Petersburg
- Spain (4):
  - Galderma Investigational Site, Barcelona
  - Galderma Investigational Site, Esplugues de Llobregat
  - Galderma Investigational site, Madrid
  - Galderma Investigational Site, Valencia
- Ukraine (6):
  - Galderma Investigational Site, Dnipropetrovsk
  - Galderma Investigational Site, Ivano-Frankivsk
  - Galderma Investigational Site, Kharkiv
  - Galderma Investigational Site, Kyiv
  - Galderma Investigational Site, Lviv
  - Galderma Investigational Site, Uzhhorod

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CD5789 (Trifarotene) 50µg/g Cream | Placebo Cream
Started | 602 | 610
Completed | 558 | 573
Not Completed | 44 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CD5789 (Trifarotene) 50µg/g Cream | Placebo Cream | Total
Number analyzed (Participants) | 602 | 610 | 1212
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 276 | 294 | 570
  Between 18 and 65 years | 326 | 316 | 642
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 357 | 338 | 695
  Male | 245 | 272 | 517
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 60 | 62 | 122
  Not Hispanic or Latino | 542 | 548 | 1090
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 2 | 6 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 27 | 42 | 69
  White | 565 | 554 | 1119
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 5 | 3 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  Romania | 64 | 65 | 129
  Hungary | 74 | 66 | 140
  United States | 124 | 154 | 278
  Czechia | 63 | 60 | 123
  Ukraine | 71 | 74 | 145
  Poland | 92 | 96 | 188
  Russia | 100 | 81 | 181
  Spain | 14 | 14 | 28
Investigator Global Asssessment [Number; unit: participants] — 0 - Clear (Clear skin with no inflammatory or non-inflammatory lesions.)
  1. - Almost Clear (A few scattered comedones and a few small papules.)
  2. - Mild (Easily recognizable; less than half the surface is involved. Some comedones and some papules and pustules.)
  3. - Moderate (More than half of the surface is involved. Many comedones, papules and pustules. One nodule may be present.)
  4. - Severe (Entire surface is involved. Covered with comedones, numerous papules and pustules. Few nodules may be present.)
  participants
    Clear | 0 | 0 | 0
    Almost Clear | 0 | 0 | 0
    Mild | 0 | 0 | 0
    Moderate | 602 | 610 | 1212
    Severe | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Investigator Global Assessment (IGA) Score of 1 (Almost Clear) or 0 (Clear)
Description: Number of subjects who achieved an Investigator Global Assessment (IGA) score of 1 (almost clear) or 0 (Clear) and at least a 2-grade improvement from Baseline to Week 12.
Time Frame: From Baseline to Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | CD5789 (Trifarotene) 50µg/g Cream | Placebo Cream
Number analyzed (Participants) | 598 | 609
Participants | 255 | 157

ADVERSE EVENTS:
Time Frame: Each participant's adverse events were collected starting at the first visit (screening) until the last visit (Week 12).
Arm/Group | CD5789 (Trifarotene) 50µg/g Cream | Placebo Cream
All-Cause Mortality (participants affected / at risk) | 0/602 | 0/610
Serious Adverse Events (participants affected / at risk) | 2/602 | 4/610
Other Adverse Events (participants affected / at risk) | 21/602 | 5/610
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CD5789 (Trifarotene) 50µg/g Cream (N=602) | Placebo Cream (N=610)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Suicide Attempt (Psychiatric disorders) | 1 | 1
Major Depression (Psychiatric disorders) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CD5789 (Trifarotene) 50µg/g Cream (N=602) | Placebo Cream (N=610)
Sunburn (Injury, poisoning and procedural complications) | 2 | 0
Drug Administered at Inappropriate Site (Injury, poisoning and procedural complications) | 1 | 0
Blood Bilirubin Increased (Investigations) | 0 | 1
Blood Creatinine Increased (Investigations) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Eyelid Exfoliation (Eye disorders) | 1 | 0
Eyelid Edema (Eye disorders) | 1 | 0
Application Site Irritation (General disorders) | 15 | 0
Application Site Puritis (General disorders) | 5 | 2
Application Site Pain (General disorders) | 4 | 0
Application Site Dryness (General disorders) | 3 | 0
Application Site Erosion (General disorders) | 1 | 0
Application Site Erythema (General disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 2 | 0
Skin Fissures (Skin and subcutaneous tissue disorders) | 1 | 0
Herpes Simplex (Infections and infestations) | 1 | 0
Tinea Versicolor (Infections and infestations) | 1 | 0
Oral Herpes (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/88/NCT02556788/Prot_001.pdf
  • Statistical Analysis Plan (2015-10-05): https://cdn.clinicaltrials.gov/large-docs/88/NCT02556788/SAP_002.pdf